CLINICAL TRIAL: NCT06454591
Title: Developing a Rapid Objective Functional MRI Assessment and Report to Characterize Functional Abilities and Predict Persistent Symptoms Following Traumatic Brain Injury
Brief Title: Rapid MRI for Assessing Functional Abilities and Predicting TBI Outcomes
Status: Recruiting | Type: Observational
Sponsor: D.J Cook (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor-Investigator, D.J Cook, Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 6041393
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TBI patients
- Individuals with chronic TBI
- Caregivers of individuals with chronic TBI
- Clinicians who treat individuals with TBI
- Legal and insurance personnel

SUMMARY:
Our project aims to develop a rapidly acquired and communicated MRI assessment and report that incorporates functional and structural imaging to convey information about functional neurological insults following traumatic brain injury (TBI) that are not typically visible on clinical imaging. Within this framework, there are two sub-studies. The first is a prospective study of patients with TBI who will have an MRI in the sub-acute period after their injury, followed by clinical assessments up to 90 days post-injury. A model will be developed to link MRI biomarkers to persistent symptoms of TBI. The second sub-study will use a focus group methodology to develop the report content and format with input from several groups of stakeholders.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) can range from mild (mTBI) to moderate and severe (msTBI), and 69 million individuals worldwide sustain a TBI annually. There are many unanswered questions related to the diagnosis of TBI, the prediction of recovery, and the selection of effective treatments. For a subset of patients with TBI, persistent symptoms (PS) can substantially reduce quality of life. Particularly for mTBI, these impairments occur frequently without evidence of structural damage to the brain on MRI or CT. The lack of objective evidence of damage can limit a patient's access to clinical resources, insurance coverage and compensation related to their injury.

Furthermore, clinicians often have difficulty predicting TBI patients' course and extent of recovery. Preliminary evidence suggests that combining several novel types of MRI techniques may enable the detection of changes in individuals with TBI and provide information about patient recovery. Therefore, our proposed research project will assess individuals with TBI using novel MRI and a battery of assessments that examine how they function (functional assessments) in the acute stages after injury with a complete reassessment of function three months after injury. These procedures will be performed in 200 patients. Overall, this project will incorporate TBI survivors, family members/caregivers, clinicians, and members of the legal/insurance community to address four goals:

1. To develop reports for survivors and their supporters to communicate MRI and functional assessment findings. This report will help survivors understand their injuries and symptoms and suggest treatments. Additionally, a more technical report will be developed for clinicians and legal/insurance personnel to support diagnosis, direct testing, and aid in choosing therapeutic approaches. Focus groups will be conducted for each group to develop the report content and format.
2. To link MRI findings to neurological function and symptoms. The use of several MRI sequences increases our ability to identify deficits. However, this large amount of information may be difficult for a clinician to review, synthesize and use to predict patient function. The investigators developed a method to summarize the MRI data into intuitive outputs to address this. These outputs are linked to function and allow clinicians and patients to connect the damage detected by MRI to impairments in function.
3. To develop a tool to assess the risk of PS 90 days after injury using MRI and clinical data collected early after injury.
4. To develop a comprehensive MRI protocol that can be performed within the shortest possible time on any clinical MRI scanner to make this testing widely accessible. For the complete MRI protocol used in this study, the total time will be 45 minutes, with five types of MRI collected. The investigators will perform analyses where one or more MRI types is removed from the analysis to understand whether all types collected are necessary to achieve the outcome. This will allow us to reduce the scan time as the clinical protocol is developed.

Findings from this work will be impactful for the following reasons: (1) the development of a report will allow patients and caregivers to be more informed about their path to recovery; (2) the development of an accessible clinical protocol and report will allow clinicians to access functional neuroimaging; (3) a protocol that links functional neuroimaging changes to functional impairment will provide evidence that injury is linked to signs/symptoms in TBI; (4) identification of patients at risk for PS combined with a comprehensive functional evaluation in the acute stages of injury will allow clinicians to focus on early therapy to prevent PS; and (5) development of the shortest possible protocol for data acquisition that increases patient comfort and increases accessibility to functional neuroimaging in the clinical setting.

ELIGIBILITY:
Sub-acute MRI study

Inclusion Criteria:

- Diagnosis of TBI

Exclusion Criteria:

* Self-reported history of brain surgery
* Self-reported history of major neurologic, psychiatric or substance use disorder
* Contraindications to MRI
* Inability to follow-up at 30 and 90 days

Focus group study Individuals with chronic TBI

Inclusion Criteria:

- Diagnosis of TBI greater than one year prior

Exclusion Criteria:

- Major neurologic, psychiatric or substance use disorder

Caregivers of individuals with chronic TBI

Inclusion Criteria:

- Relation who was diagnosed with TBI greater than one year prior that individual was the primary caregiver for

Exclusion Criteria:

- Major neurologic, psychiatric or substance use disorder

Clinicians who treat TBI

Inclusion Criteria:

- Employment as a physician or allied health professional who has spent greater than 50% of their time treating TBI patients for at least two years of their career

Exclusion Criteria:

-N/A

Inclusion Criteria:

- Employment as a personal injury lawyer or insurance adjuster who has spent greater than 50% of their time on TBI cases for at least two years of their career

Exclusion Criteria:

-N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sub-acute MRI study Individuals with mTBI within previous 7 days and individuals with moderate or severe TBI in previous 90 days
  Focus group study Individuals with chronic TBI Caregivers of individuals with chronic TBI Clinicians who treat TBI Legal and insurance personnel who handle TBI cases
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Model performance for prediction of post-concussion symptom scale (PCSS) score | Model predicts 90-day PCSS score
  R-squared and mean absolute error for model performance for mild TBI and moderate/severe TBI models

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Cook, MD, PhD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Queen's University, Kingston, Ontario